CLINICAL TRIAL: NCT04320654
Title: Will Patients With Low Back Pain Benefit From the Advice of Staying Active
Brief Title: Advice of Staying Active for Sub Acute Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Khaled Shoukry, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5402
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: different groups each will receive specific intervention at the same time
Who Masked: Participant
Masking Description: sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- advice of staying active (Experimental): The patients will be advised to stay as physically active as possible and continue their everyday activities as normally as possible.
  Interventions: Other: exercise
- walking program (Experimental): Patients will be encouraged to go about their normal daily activities. At week one, patients will be asked to familiarize themselves with wearing the pedometer and recording their daily steps in a walking diary for the subsequent 7 days. The patients will return to see the physiotherapist at the end of week one to discuss any issues with the program, pedometer or recording of desired information. A step target for week two will be agreed between the physiotherapist and the patient by referring to the mean daily step count recorded at baseline, and the average step count calculated from the walking diary
  Interventions: Other: exercise
- Backward walking (Experimental): All patients will be instructed to walk at their desired pace 3 days per week with a steady rhythm. The duration of each training session will initially be 15 minutes and will gradually increase, and finally reach 25 minutes, for every session (Hao Chen, 2011). There will be no constraint or indication about head and trunk position during backward training
  Interventions: Other: exercise
- Targeted home-based hip exercise (Experimental): Patients who will be assigned in this group will perform a hip exercise program for six weeks, three times / week to ensure an adequate recovery between exercise sessions (appendix V). The strengthening exercises will focus on strengthening the gluteus maximus (GMax), gluteus medius (GMed), gluteus minimus (GMin) and short hip external rotator muscles (Distefano et al., 2009).
  Interventions: Other: exercise
- control group (No Intervention): The patients will not be given any intervention and will be asked to come after 6 weeks for re-assessment

INTERVENTIONS:
Other: exercise — The aim of this intervention is to increase patients average daily step count. The walking program is a behavior change intervention in which the pedometer will be used as a tool to help the patients monitor their activity levels.
  Arms: Backward walking; Targeted home-based hip exercise; advice of staying active; walking program

SUMMARY:
The variabilities in the management approaches for patients with LBP reflect uncertainty about the optimal approach. Therefore, there is a need for the implementation of early treatment strategies relying on an evidence-based knowledge to treat the problems and reduce the risk for recurrence and chronicity of LBP.

Advice is considered as the 'first in line' for the treatment of patients with LBP and is recommended in all international guidelines, yet it is under-utilized by the general practitioners. The current evidence in favor for the advice of staying active for patients with LBP is limited, with small or no benefits in pain relief, functional improvement or sick leave compared to rest in bed. Consequently, there is a huge gap between the evidence and practice.

So, the current study aimed at filling this gap and expanding the previous findings by investigating the effect of the advice of staying active on the level of perceived pain, physical activity level, postural control and functional disability in patients with low risk LBP (with a total score of three or less based on the STarT Back Tool score).

DETAILED DESCRIPTION:
In spite of the great effort, LBP remains a significant burden on the society and can cause a disturbing impact on the functional ability during the productive years of the individuals. It is important to find pragmatic treatments that not only reduce the pain, but also decrease the disability. Activity monitoring in real life has the potential to change our concept of outcomes, and as a result, expand our ideas about the appropriateness of the interventions in rehabilitation.

The international guidelines vary but agree on advising patients with LBP to remain physically active. The National Institute for Clinical Excellence (NICE)'s updated guideline on the LBP recommends encouraging people to continue with their normal activities as far as possible. NICE found that there were no randomized controlled trials (RCTs) (which are the best way of investigating the efficacy of a treatment) that compared the effect of the advice of staying active with no advice or the advice to rest.

Despite the guidelines, it was reported that many health care providers are still too restrictive and believe that LBP requires some avoidance of activities and to remain off- work. Many general practitioners do not give advice on daily activities to patients with back pain and there is confusion about what constitutes an effective advice. Only 12% of the physiotherapists identify correctly the guidelines, and most of them do not agree with these guidelines regarding the return to work or activity. Investigating the benefit of the advice of staying active and different active intervention programs in patients with low risk NSLBP may help in developing recommendations for the physiotherapists responsible for reviewing exercise protocols for patients with LBP.

Therefore, the improvement of the primary care management of patients with LBP has the potential to reduce the long-term effects of back pain, including persistent disabling symptoms, low quality of life, and reduced capacity to work. The advice of staying active may not only be a treatment to improve the recovery from LBP, but also an opportunity to promote physical activity for other health benefits, such as improved cardio-metabolic function, blood pressure, and reduced body fatness.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are between 18 - 65 years of age
* able to stand and walk without assistance.
* Patients will also be included if they have a history of non specific low back pain classified as low risk of poor outcome with a total score of three or less based on the STarT Back Tool score (Hill et al., 2008).
* The back-pain episode is subacute

Exclusion Criteria:

* Patients will be excluded if they have any neurological disease or balance deficits due to vestibular disorders, such as vertebrobasilar insufficiency and visual disorders,
* systemic infection,
* current pregnancy,
* severe musculoskeletal deformity (scoliosis or kyphosis),
* injury to the lower extremity that would interfere with testing or a history of any surgery in the three months prior to testing.
* Patients will also be excluded if they have pain below the knee consistent with a disc herniation, presence of neurological signs, serious spinal complications (e.g., vertebral fracture, tumor or infection),
* spinal stenosis,
* confounding conditions such as extreme obesity, severe scoliosis, significant anatomical leg length inequality, previous spinal surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
level of perceived pain by Visual analogue scale | six weeks
  The Visual analogue scale will be used for measuring the pain intensity the scale ranges from 0 to 10 where 0 means no pain and 10 means severe intolerable pain.

SECONDARY OUTCOMES:
number of steps | six weeks
  A spring-leverd pedometer (Yamax Digiwalker CW-701, Yamax, Japan) will be used to assess the number of steps. The number of steps will be used as an indicator for the level of physical activity

IPD SHARING:
Plan to Share IPD: No